CLINICAL TRIAL: NCT00002655
Title: Cryosurgical Destruction of Surgically Incurable Liver Tumors
Brief Title: Cryosurgery in Treating Patients With Liver Cancer or Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 93-0092.cc; NCI-V95-0657 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cryosurgery

SUMMARY:
RATIONALE: Cryosurgery kills cancer cells by freezing them during surgery.

PURPOSE: Phase I/II trial to study the effectiveness of cryosurgery in treating patients with unresectable primary liver cancer or liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety and efficacy of liquid nitrogen necrosis of liver lesions using a commercially available intraoperative cryosurgical system, with placement of the cryoprobe and subsequent monitoring by high-resolution ultrasound. II. Use this technique on selected patients with surgically unresectable metastatic or primary liver cancer whose disease appears confined to the liver and who are potentially curable if all tumor in the liver can be destroyed. III. Quantitate the quality and duration of survival, identify recurrence of hepatic malignant disease, and identify any morbidity from the procedure.

OUTLINE: Cryosurgery. Liquid nitrogen freezing of tumor using a cryoprobe placed and maintained under ultrasound guidance.

PROJECTED ACCRUAL: 50 patients will be treated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven metastatic or primary malignant disease of the liver No extrahepatic regional or distant metastases No primary tumors commonly associated with local spread or metastases to other sites, e.g.: Gastric cancer Pancreatic cancer Breast cancer Lung cancer Liver lesions considered unresectable because of location in relation to major vascular structures or involvement of multiple hepatic segments Tumor extent and location such that cryosurgery expected to destroy all tumor and render patient disease-free Tumor volume no greater than 50% of total hepatic volume on CT No more than 12 lesions

PATIENT CHARACTERISTICS: Age: Over 21 Other: Overall health permitting safe laparotomy Blood/body fluid analyses and imaging/exams for tumor measurement within 1 month prior to registration

PRIOR CONCURRENT THERAPY: Prior liver resection, radiotherapy, or chemotherapy allowed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-03; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg V. Stiegmann, MD, Study Chair — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Denver, Colorado, United States